CLINICAL TRIAL: NCT05860881
Title: A Randomised Double-blind Placebo-controlled Trial of Topical Sirolimus in Chemoprevention of Facial Squamous Cell Carcinomas in Solid Organ Transplant Recipients
Brief Title: Topical Sirolimus in Chemoprevention of Facial Squamous Cell Carcinomas in Solid Organ Transplant Recipients (SiroSkin)
Acronym: SiroSkin
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Melanoma and Skin Cancer Trials Limited (Other)
Collaborators: Monash University (Other); The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 01.21 SiroSkin
Record Dates: First submitted 2023-05-08; First posted 2023-05-16 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Solid Organ Transplant Recipients; Skin Cancer
MeSH Terms: conditions — Skin Neoplasms | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical Sirolimus (Experimental): Topical 1% sirolimus cream applied daily to the face for 24 weeks
  Interventions: Drug: Sirolimus Topical Cream
- Placebo (Placebo Comparator): Topical placebo cream applied daily to the face for 24 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sirolimus Topical Cream — The intervention topical cream consists of sirolimus 1% in a vehicle. Patients randomised to the intervention will be required to apply the sirolimus topical cream to their face for 6 months
  Other Names: Rapamycin
  Arms: Topical Sirolimus
Other: Placebo — Cream containing only the base, or vehicle.
  Other Names: Vehicle alone
  Arms: Placebo

SUMMARY:
01.21 SiroSkin is a phase 3, double-blind, multi-centre, parallel-arm, randomised, placebo-controlled trial to evaluate the use of topical 1% sirolimus in the chemoprevention of skin cancer, versus placebo, applied every night for 24 weeks in solid organ transplant recipients.

DETAILED DESCRIPTION:
Keratinocyte carcinomas are a major burden affecting mortality and morbidity in solid organ transplant recipients (SOTRs). Due to an increased prevalence of skin cancers, SOTRs require recurrent skin checks and frequent skin cancer surgery. The gold standard of treatment is surgery, enabling complete remission and a cure in the majority of cases. Despite this, there is no effective way of preventing new cancers from developing in the same area.

Oral sirolimus is a selective immunosuppressant agent which has proven to reduce the burden of skin cancer; however, it is poorly tolerated due to side effects. Topical sirolimus has proven effective in reducing the skin cancer burden in animal models and is safe on the face of patients with tuberous sclerosis. An initial 12-week phase II clinical trial recently conducted by the research team suggested topical sirolimus to be safe and effective, as it reduced the early signs of skin cancer without any major side effects.

In this phase III randomised, double-blind, placebo-controlled study, we propose using 1% topical sirolimus applied to the face on a regular basis for 24 weeks. We aim to determine whether this topical cream can fill a major gap in our current therapies by reducing the onset of new skin cancers and therefore reduce the burden of disease in terms of number of biopsies and surgeries, and potential hospitalisations and death.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged 18 years or older and able to provide consent
2. Have received an organ transplant equal to or greater than 12 months prior to consent
3. Have had at least 1 SCC/BCC in the past 5 years
4. Have at least 5 keratotic lesions on their face at inclusion or have a history of keratinocyte cancer on the face in the past 5 years

Exclusion Criteria:

1. Are currently receiving sirolimus or everolimus orally*
2. Have a skin cancer on their face requiring excisional surgery**
3. Have an open wound on their face requiring treatment
4. Are pregnant or planning to become pregnant in the next 6 months
5. Anticipate elective medical events which may prevent daily cream application.
6. Are unable to provide informed consent, complete questionnaires and attend trial site for visits
7. Are participating in another clinical trial with an investigational drug/device aiming to reduce skin cancers or affect level of immunosuppression
8. Planning to move overseas within 2 years

(*)Patients are eligible to join the study after ceasing treatment and after a washout period of 16 days for sirolimus and 8 days for everolimus.

(**) Once treatment of the lesion is completed these patients can be re-screened.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 7 days (168 hours) prior to their baseline & screening visit (D0) and agree to use adequate methods of contraception for the duration of drug administration.
Enrollment: 146 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
KC development | 2 years
  The number of keratinocyte carcinomas (KCs) on the treated area compared with placebo, at the completion of 24 weeks of topical 1% sirolimus then at 12 and 24 months.

SECONDARY OUTCOMES:
The occurrence of KCs | 2 years
  The occurrence of keratinocyte carcinomas (KCs) on the treated area at the completion of 24 weeks of topical 1% sirolimus then at 12 and 24 months follow up.
The number of biopsy-proven SCCs | 2 years
  The number of biopsy-proven squamous cell carcinomas (SCCs) at the completion of 24 weeks of topical 1% sirolimus, then at 12 and 24 months follow up on the treated area.
The occurrence of biopsy-proven squamous cell carcinomas (SCCs) | 2 years
  The occurrence of biopsy-proven squamous cell carcinomas (SCCs) at the completion of 24 weeks of topical 1% sirolimus, then at 12 and 24 months follow up on the treated area.
The number of IECs, BCCs and subtypes of SCCs or BCCs | 2 years
  The number of intraepidermal carcinomas (IECs), basal cell carcinomas (BCCs) and subtypes of squamous cell carcinomas (SCCs) or BCCs at each of the aforementioned time-points on the treated area.
The occurrence of IECs, BCCs and subtypes of SCCs or BCCs | 2 years
  The occurrence of intraepidermal carcinomas (IECs), BCCs and subtypes of squamous cell carcinomas (SCCs) or basal cell carcinomas (BCCs) at each of the aforementioned time-points on the treated area.
The number of AKs | 2 years
  The number of facial actinic keratosis of each patient at recruitment compared to 3, 6, 12 and 24 months on photographic images and counts.
Cost-effectiveness | 2 years
  The cost-effectiveness of utilising topical sirolimus therapy on SOTRs in comparison to the current standard of care, being surgical intervention, in the management of KCs.
The number and occurrence of intervention-related side effects | Up to 30 days post end of treatment
  The number and occurrence of intervention-related side effects by reviewing any Urgent Safety Measures (USMs), Suspected Unexpected Serious Adverse Reaction (SUSARs), Serious Adverse events (SAEs) and skin-related AEs occurring up to 30 days post-EOT. Adverse events will be reviewed by type, grade according to CTCAE v5.0 and relatedness to treatment.
Compliance | 6 months
  The feasibility of the 1% sirolimus treatment in SORTs by reviewing completion of the 24-week application course and the total number of doses applied during the course.
Quality of life (EQ-5D-5L) | 2 years
  To evaluate the participants' experience by monitoring side effects and issuing participant surveys such as the EuroQol 5-dimensional (EQ-5D-5L) questionnaire.The EQ-5D-5L questionnaire is a preference-based measure of health status - commonly used in trial-based economic evaluation and is suited for cancer-specific instruments. This tool contains 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The scoring algorithm for the EQ-5D-5L will use the Australian-based value set resulting in scores between 0 and 1 (1 meaning full health).
Quality of life (BaSQoL) | 2 years
  Quality of life will also be assessed with the Basal and Squamous Cell Carcinoma Quality of Life (BaSQoL) questionnaire which covers the experiences of skin cancer treatment, diagnosis-related issues and long-term behavioural changes. There are 16 questions and 5 domains including: behaviours, diagnosis and treatment, worries, appearance, and other people. Each question is scored from 0 to 3 with 0 indicating no impact and 3 indicating strong impact on quality of life. The mean scores for each domain are calculated however, the BaSQoL has no summary score or index. The lower the score the lower the impact of the cancer on the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Kiarash Khosrotehrani, MD PhD FACD, Study Chair — The University of Queensland
Locations (6):
- Australia (6):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Skin Health Institute, Carlton, Victoria
  - The Alfred Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dousset L, Chambers DC, Webster A, Isbel N, Campbell S, Duarte C, Collins L, Damian D, Tseng A, Karlsen E, Ilinsky OV, Brown S, Schaider H, Soyer HP, Ospino DA, Hogarth S, Chong AH, Mar V, McKenzie S, Gin D, Fernandez-Penas P, Kern JS, Loewe K, Roy E, Herschtal A, Khosrotehrani K. Trial protocol for SiroSkin: a randomised double-blind placebo-controlled trial of topical sirolimus in chemoprevention of facial squamous cell carcinomas in solid organ transplant recipients. Trials. 2024 Nov 22;25(1):789. doi: 10.1186/s13063-024-08619-3. PMID 39578921
- See also: Detailed information on the SiroSkin trial — https://www.masc.org.au/siroskin/